CLINICAL TRIAL: NCT04683757
Title: A Prospective Cohort Study： the Establishment of a Survival Prediction Model for ER Positive / HER-2 Negative Advanced Breast Cancer
Brief Title: The Establishment of a Survival Prediction Model for ER Positive / HER-2 Negative Advanced Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ying Wang (Other)
Responsible Party: Sponsor-Investigator, Ying Wang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Other Study IDs: 2017-KY-19
Record Dates: First submitted 2020-12-19; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; a Survival Prediction Model
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The target of this study is to detect the gene mutation of tumor tissue or peripheral blood circulation tumor DNA of tumor patients. 10ml of tissue or fresh peripheral blood should be collected as the test sample and stored at room temperature. On the same day, it was sent to the "cell and molecular diagnosis center" of our hospital for DNA isolation and extraction, secondary sequencing, and detection of related biomarkers, such as erbB2 / TP53 / PIK3CA / ErbB4 / CCND1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Establishment of a Survival Prediction Model — a nomogram to predict the survival of patients with ER positive / HER-2 negative advanced breast cancer

SUMMARY:
This project is a prospective, clinical cohort study initiated by researchers to study the high-risk factors affecting the overall survival of newly diagnosed ER + / HER2 - advanced breast cancer patients and to establish a prediction model of ER + / HER2 - advanced breast cancer patients affecting overall survival. This project is the first prospective prediction model for the survival of patients with advanced breast cancer, and it is also the first time to establish a survival prediction model for ER-positive / HER2 negative advanced breast cancer suitable for China's national conditions. According to the survival outcome predicted by the model, the newly diagnosed ER positive / HER2 negative advanced breast cancer was divided into three groups: low, medium, and high risk, which provided an important theoretical basis for further design of randomized controlled clinical research and guidance of individualized precise treatment scheme for different groups in the future.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing the informed consent form, 18 years old ≤ 70 years old, female
2. ER positive breast cancer confirmed by pathology: ER positive (≥ 1%) by immunohistochemistry
3. Newly diagnosed advanced patients, including patients with early breast cancer who have evidence of recurrence and metastasis after adjuvant therapy and patients with stage IV breast cancer at the first visit
4. Patients who are willing to receive follow-up treatment in the research center.

Exclusion Criteria:

1. ErbB-2 gene amplification was recorded by fish (defined as HER2 / CEP17 ratio ≥ 2) or chromogenic in situ hybridization (CISH) or IHC (defined as ihc3 +, or ihc2 + confirmed by fish or CISH) was used to record HER2 positive tumors.
2. Any form of anti-cancer treatment has been carried out for recurrent or metastatic lesions
3. Combined with other malignant tumors or had other malignant tumors in recent 5 years
4. Patients with nervous system disorders caused by diseases or obvious mental disorders will affect patients' right to know, compliance or make them in a dangerous state
5. Patients with life expectancy less than 3 months

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer
Sampling Method: Probability Sample
Enrollment: 288 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
overall survival，OS | 5 years
  The time from the beginning of treatment to the death of the patient
Tumor specific survival time, CSS | 5 years
  The follow-up started from the first day of confirmed recurrence and metastasis. The end point of follow-up was the death caused by tumor related causes.

SECONDARY OUTCOMES:
Progression Free Survival，PFS | 2 years
  The time from the beginning of treatment to the progression or death of the patient.
5-year survival rate | 5 years
  the survival rate in 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat Sen Memorial Hospital，Sun Yat sen University, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital， Sun Yat-sen University, Guanzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No